CLINICAL TRIAL: NCT01734304
Title: Active Immunotherapy of Patients With Acute Myeloid Leukemia Using Autologous Dendritic Cells Transfected With RNA Encoding Leukemia-associated Antigens
Brief Title: DC Vaccination for Postremission Therapy in AML
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, PD Dr. Marion Subklewe, Prof. Dr. med. Marion Subklewe, Ludwig-Maximilians - University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-022446-24
Record Dates: First submitted 2012-10-17; First posted 2012-11-27 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: vaccination; postremission therapy; acute myeloid leukemia; dendritic cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DC vaccination (Experimental): Vaccination with TLR7/8-matured DCs electroporated with mRNA encoding WT1, PRAME, and CMVpp65
  Interventions: Biological: DC vaccination for postremission therapy in AML

INTERVENTIONS:
Biological: DC vaccination for postremission therapy in AML — Vaccination with TLR7/8-matured DCs electroporated with mRNA encoding WT1, PRAME, and CMVpp65

SUMMARY:
The aim of this study is to determine the feasibility and safety of an autologous DC immunotherapy in patients with AML of non-favorable risk profile.

DETAILED DESCRIPTION:
Patients ≥ 18 years of either gender with AML of non-favorable risk profile in CR or CRi not being eligible for allogeneic stem cell transplantation will receive as intradermal injections at two different sites up to ten immunotherapies with autologous DCs presenting two leukemia-associated antigens and one CMV antigen conserved in cryomedium over a time span of 26 weeks. Phase I will test the safety and toxicity in a small group of patients (n=6). After at least four vaccinations of three patients, the safety and toxicity data will be presented to the Data safety monitoring board (DSMB). Only after the DSMB has no objectives against the continuation of the trial, further patients will be included into the trial. Again, after three more patients, receiving a minimum of four vaccines, clinical data will be presented to the DSMB, and phase I will be terminated. The decision for continuation of the trial will be done by the DSMB. If there are no objectives by the DSMB, the trial will continue and evaluation will be started in a larger group of patients (n=14). During the phase II trial, safety and toxicity will be evaluated in a larger co-hort of patients). Besides, preliminary assessment of efficacy will be performed including induction of immunological responses to leukemia associated antigens as well as to a viral antigen (CMV), MRD control, time to progression of disease and ECOG performance status.

ELIGIBILITY:
Inclusion Criteria:

* Patients male or female, age ≥ 18 years, biological age ≤ 75 years
* Patients with AML of non-favorable risk profile or with AML and sole NPM1 mutation and confirmed increase of MRD load as detected by RQ-PCR (in two measurements at least four weeks apart)
* CR or CRi after intensive induction chemotherapy (TAD, HAM, sHAM, 3+7 anthracycline + cytarabine regimen, or equivalent)
* Negative HIV test, negative hepatitis B and C test
* Negative pregnancy test in women of childbearing potential
* Ability to understand and willingness to sign a written informed consent

Exclusion Criteria:

* Patients suitable for allogeneic HSCT (indication for allogeneic HSCT, adequate donor, no contraindication for allogeneic HSCT)
* Patients with AML with favorable risk profile:
* APL (AML M3)
* inv(16), t(16;16), or del(16) as sole anomaly
* t(8;21) as sole anomaly
* biallelic CEBPA mutation as sole anomaly
* NPM1 mutation as sole anomaly, unless with confirmed increase of MRD load
* Prior allogeneic HSCT
* Anemia (Hb < 9,0 mg/dl)
* Leukopenia (< 4,0 G/l)
* Transfusion refractory thrombocytopenia (< 30 G/l platelets despite adequate number of transfusions)
* Active clinically relevant autoimmune disease
* Active immunodeficiency syndromes
* Known allergy to GM-CSF, TNF, IFN-γ, IL-4, IL-1 beta, PGE2, R848, Human AB Serum, DMSO, HSA
* Continuous therapy with corticosteroids or other immunosuppressive drugs during the trial
* Present substance abuse or any other factor that could limit the subject's ability to comply with study procedures
* Severe organ dysfunction:
* Creatinine > 2,5 mg/ml
* Bilirubin > 3,0 mg/ml
* ALAT and ASAT > 3 x upper normal limit
* Respiratory insufficiency with pO2 < 60 mmHg
* Clinically relevant coronary heart disease of ventricular arrhythmia, congestive heart failure > grade II NYHA
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study
* Simultaneous participation in another clinical trial or participation in any clinical trial involving an investigational medicinal product within 30 days prior to written informed consent for this trial

Exclusion criteria regarding special restrictions for females:

* Current or planned pregnancy or nursing women
* Females of childbearing potential, who are not using and not willing to use medically reliable methods of contraception for the entire study duration and at least 3 months thereafter (such as oral, injectable, or im-plantable contraceptives, or intrauterine contraceptive devices) unless they are surgically sterilized/hysterectomized or there are any other criteria considered sufficiently reliable by the investigator in individual cases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
% of grade I/II and grade III/IV toxicities | 30 weeks

SECONDARY OUTCOMES:
Immune responses to applied antigens | 30 weeks
Control of minimal residual disease | 30 weeks
Time to progression of disease | 30 weeks
ECOG performance status | 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marion Subklewe, PD Dr, Principal Investigator — Department of Medicine III; Hospital of the University of Munich,
Locations (1):
- Hospital of the University of Munich, LMU; Department od Medicine III, Munich, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lichtenegger FS, Schnorfeil FM, Rothe M, Deiser K, Altmann T, Bucklein VL, Kohnke T, Augsberger C, Konstandin NP, Spiekermann K, Moosmann A, Boehm S, Boxberg M, Heemskerk MH, Goerlich D, Wittmann G, Wagner B, Hiddemann W, Schendel DJ, Kvalheim G, Bigalke I, Subklewe M. Toll-like receptor 7/8-matured RNA-transduced dendritic cells as post-remission therapy in acute myeloid leukaemia: results of a phase I trial. Clin Transl Immunology. 2020 Mar 3;9(3):e1117. doi: 10.1002/cti2.1117. eCollection 2020. PMID 32153780